CLINICAL TRIAL: NCT03162185
Title: The Effects of Serotonergic Challenge on Motor Learning and Neuroplasticity
Brief Title: Serotonin and Motor Plasticity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MaxPlanckHCBS
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Healthy Controls
Keywords: Neuroplasticity; SSRI; Motor Learning
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Half of the participants (n = 30) will receive 20mg of the SSRI Escitalopram.
  Interventions: Drug: Escitalopram
- Control group (Placebo Comparator): Half of the participants ( n= 30) will receive the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Experimental group participants (n = 30) will receive 20 mg of Escitalopram for 7 days.
  Arms: Interventional group
Drug: Placebo — Control group participants (n = 30) will receive a placebo for 7 days.
  Arms: Control group

SUMMARY:
With this study, the investigators aim to test whether acute administration of selective serotonin reuptake inhibitors (SSRI) improves motor performance in a sequential motor learning task in comparison to placebo in healthy humans.

DETAILED DESCRIPTION:
Microdialysis findings in animal models provide evidence for a monoaminergic augmentation of motor function. However, this evidence is largely limited to noradrenaline and dopamine, with little evidence to support a similar effect for serotonin. What remains to be tested therefore, is whether acute serotonergic administration induces neural or behavioral changes during motor learning also. Using a sample of 60 female participants (with the possible inclusion of male participants at a later date), the investigators aim to test the effects of a serotonergic challenge on motor learning and plasticity in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* female
* right-handed
* healthy
* has taken oral contraceptives (ovulation inhibitor) continuously for at least 3 months
* has read and agreed to study parameters

Exclusion Criteria:

* tattoos on head or neck
* non-removable metal on or in body
* alcohol abuse
* is currently taking medication
* smokes more than 3 cigarettes per day
* positive drug test
* pregnancy
* plays an instrument professionally
* plays videogames more than 2 hours per week
* is a professional athlete
* suffers from migraines
* has taken part in another study, where motor learning skills and/or medication is a factor, in the last 3 months
* heart rhythm disorders (long QT)
* hypertension
* calcium or magnesium deficiency
* neurological disorders
* chronic metabolic disorders
* liver or kidney diseases
* immunodeficiency
* endocrine disorders
* psychiatric disorders
* tumors
* injuries to the head and brain

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Pinch Force Task. | 1 week
  The primary outcome measure will be reaction time and accuracy of motor responses, as measured by the Pinch Force Task. This will be applied to both the experimental (SSRI) and control (Placebo) groups.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Villringer, Study Chair — Max Planck Institute for Human Cognitive and Brain Sciences; Julia Sacher, Study Director — Max Planck Institute for Human Cognitive and Brain Sciences
Locations (1):
- Max Planck Institute for Cognition and Brain Sciences, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No